CLINICAL TRIAL: NCT00505453
Title: A Phase III, Open-Label, Single-Dose Study to Evaluate the Safety and Immunogenicity of Fluviral® Trivalent Split Virion Influenza Vaccine (2007 - 2008 Season) in Adults Ranging in Age From 18 to 60 Years and 61 Years and Over
Brief Title: A Phase III, Open-Label, Single-Dose Study to Evaluate the Safety and Immunogenicity of Fluviral® Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110502
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Fluviral®

SUMMARY:
Vaccination is currently the most effective means of controlling influenza and preventing its complications and mortality in persons at risk.

Once a year, a meeting of WHO experts takes place, leading to a recommendation on the influenza A and B strains that should be used for the production of vaccine for the coming influenza season.

This study is designed to test the safety/reactogenicity and the immunogenicity of the Fluviral Trivalent Split Virion Influenza Vaccine containing the influenza strains recommended for the 2007-2008 season.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults, 18 years of age and older.
* Female subject of non-childbearing potential. Written informed consent obtained from subject.

Exclusion Criteria:

* Acute disease at the time of enrollment.
* Blood pressure abnormalities.
* Any immunosuppressive condition, such as HIV or cancer.
* Renal impairment, hepatic dysfunction, complicated insulin-dependent diabetes mellitus.
* Unstable cardiopulmonary disease requiring chronic medical therapy or associated with functional impairment.
* Any demyelinating disease, including Guillain-Barré syndrome.
* Alcohol consumption and/or drug abuse.
* Receipt of an influenza vaccine within 9 months prior to enrollment or of any vaccines within 30 days prior to enrollment.
* Any known or suspected allergy to the Fluviral vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2007-07; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of Fluviral influenza vaccine in adults 18 years or older | 21 days after vaccination

SECONDARY OUTCOMES:
Evaluate safety & reactogenicity: Solicited AEs | 4 days
Evaluate safety & reactogenicity: Unsolicited AEs | 21 days
Evaluate safety & reactogenicity: SAEs | entire study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Canada (2):
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 110502 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110502 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110502 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110502 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110502 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110502 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110502 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register